CLINICAL TRIAL: NCT02635529
Title: A Clinical and Radiographic Evaluation of DFDBA (Demineralised Freeze Dried Bone Allograft) With Amniotic Membrane (AM) in the Treatment of Periodontal Osseous Defects-12 Month Randomized Controlled Clinical Trial
Brief Title: DFDBA and Amniotic Membrane in the Treatment of Periodontal Osseous Defects
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_44443
Record Dates: First submitted 2015-12-07; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Periodontal Intrabony Defects

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OFD + DFDBA (Active Comparator): Intrabony defects treatment was carried out with OFD + DFDBA
  Interventions: Procedure: OFD+ DFDBA
- OFD+DFDBA+AM (Active Comparator): Intrabony defects treatment was carried out with OFD + DFDBA+ AM
  Interventions: Procedure: OFD+ DFDBA+ AM

INTERVENTIONS:
Procedure: OFD+ DFDBA — After Phase I therapy, patient's were assigned for OFD+DFDBA group. Mucoperiosteal flap were reflected.After Open Flap Debridement (OFD), DFDBA graft was placed for the treatment of intrabony defects.
  Arms: OFD + DFDBA
Procedure: OFD+ DFDBA+ AM — After Phase I therapy, patient's were assigned for OFD+DFDBA + AM group. Mucoperiosteal flap were reflected. After Open Flap Debridement (OFD). DFDBA and AM was placed for the treatment of intrabony defects.
  Arms: OFD+DFDBA+AM

SUMMARY:
Amniotic membrane may be considered as a biologically active scaffold, which in combination with Bone Replacement Grafts (BRG) can be widely used to reconstruct periodontal Intrabony Defects (IBDs), due to the presence of stem cells and growth factors. The goal of the present study was to evaluate if a biologic AM in combination with DFDBA applied in periodontal IBDs would enhance the regeneration of periodontium.

DETAILED DESCRIPTION:
Periodontitis is a bacterially induced inflammatory disease of the supporting tissues of the teeth. It is one of the major dental diseases that affect human populations worldwide and has a huge economic impact on national health care systems.The consequence of periodontitis is commonly the formation of intrabony defects.Intrabony defects are more amenable for regenerative procedures. Periodontal regeneration remains a fundamental therapeutic goal for the preservation of teeth through the restoration of health, function, and esthetics of the periodontium. Several treatment procedures like open flap debridement (OFD), autogenous bone replacement bone grafts (BRG), guided tissue regeneration (GTR), bioactive agents like EMD, rhPDGF-BB, laser assisted regeneration (LAR) have shown histologic proof of principle that the periodontal ligament apparatus can be regenerated in human studies. Intrabony defects with the depth of >3 mm and radiographic defect angle ≤ 25 are amenable for periodontal regeneration. DFDBA has stood the test of time and has shown consistent good quality patient oriented evidence in achieving periodontal regeneration with long term stability. GTR techniques have shown added advantage of space maintenance, clot stability, guided cell population, epithelial cell occlusion and the combination therapies. Periodontal regeneration with GTR and BRG demonstrates better results as compared with GTR alone. More recently in the realm of reconstructive biology, the concept of Tissue engineering (TE) has been introduced which utilizes mechanical, cellular or biologic mediators to facilitate reconstruction/regeneration of a particular tissue.

The combination of this novel biologic membrane AM and the already established BRG-DFDBA can be an added advantage in treatment of IBDs. To the best of the investigators knowledge only one clinical trial reports this combination therapy in the scientific literature. There is a need for further research in this area.

ELIGIBILITY:
Inclusion criteria:

* Age group of 25-45 years
* Moderate periodontitis with pocket probing depth more than 6mm
* Bilaterally similar intrabony defects
* Systemically healthy patients
* Vital or endodontically treated teeth
* Good compliance

Exclusion criteria:

* Medically compromised
* Pregnant and lactating women
* Smoking
* Teeth with mobility and furcation involvement

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | 1 year
  Clinical attachment level measured in mm from cementoenamel junction to base of the pocket)

SECONDARY OUTCOMES:
Plaque index | 1 year
  Plaque index is measured for periodontal health
Gingival index | 1 year
  Gingival index is measured for periodontal health
Bleeding index | 1 year
  Bleeding index is measured for periodontal health
Pocket Probing depth | 1 year
  Pocket probing depth level measured in mm from gingival margin to base of the pocket)
Bone Fill | 1 year
  Bone fill measured in mm in radiographs from alveolar crest to base of the pocket

CONTACTS AND LOCATIONS:
Overall Officials: DR JOANN P GEORGE, MDS, Study Director — Krishnadevaraya college of dental science and hospital
Locations (1):
- Krishnadevaraya college of dental sciences and hospital, Bangalore, Karnataka, India

REFERENCES:
- [Background] Kiany F, Moloudi F. Amnion membrane as a novel barrier in the treatment of intrabony defects: a controlled clinical trial. Int J Oral Maxillofac Implants. 2015 May-Jun;30(3):639-47. doi: 10.11607/jomi.3590. PMID 26009915
- See also: reference article — http://www.ncbi.nlm.nih.gov/pubmed/?term=kiany+intrabony